CLINICAL TRIAL: NCT00914147
Title: Pulmonary Function Tests (PFT) in a Phase I Patient Population
Brief Title: Lung Function Testing in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anthony F. Shields, MD PhD, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000642265; P30CA022453 (NIH); WSU-2009-004
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2020-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pulmonary Function Test (PFT) (Other): After signing consent, patients will undergo a complete spirometry test, lung volumes and diffusing capacity (DLCO) measurement utilizing the single-breath breath holding technique, according to the ATS/ERS consensus and standardization. PFT measurements will be reported as absolute values (e.g. liters) and percentage of predicted. The predicted normal values will be calculated according to sex, age, height and race using the Third National Health and Nutrition Examination Survey (NHANES III) reference equation. Predicted values for diffusion capacity will be calculated using the Morris/Polgar equation. DLCO values will be adjusted to anemia (hemoglobin levels)
  Interventions: Procedure: pulmonary function testing

INTERVENTIONS:
Procedure: pulmonary function testing — After signing consent, patients will undergo a complete spirometry test, lung volumes and diffusing capacity (DLCO) measurement utilizing the single-breath breath holding technique, according to the ATS/ERS consensus and standardization.
  Other Names: PFT

SUMMARY:
RATIONALE: Measuring how well the lungs work in patients with cancer may help doctors predict how patients will respond to treatment and help plan the best treatment.

PURPOSE: This clinical trial is studying lung function testing in patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To obtain the distribution of DLCO, FVC, and FEV_1 by pulmonary function testing (PFT) in patients with heavily pretreated locally advanced or metastatic solid tumors referred to the Karmanos Cancer Institute (KCI) Phase I Clinical Trials Program.
* To estimate the mean DLCO to within 4 units (% of predicted) of the true mean with 95% confidence.

Secondary

* To estimate the percentage of patients who meet the defined eligibility criteria (including PFT levels, especially DLCO) from the entire population enrolled in the KCI Phase I Clinical Trials Program.

OUTLINE: Patients undergo pulmonary function testing comprising spirometry test, lung volumes, and DLCO measurement utilizing the single-breath breath-holding technique. Patients then proceed to treatment on a phase I clinical trial.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Locally advanced or metastatic disease
* Disease progressed on or after standard therapy OR there is no standard therapy for the malignancy

  * Standard therapy is defined as first- or second-line therapy that has been shown to provide clinical benefit
* Life-long non-smoker
* No lung metastasis and/or pleural effusion causing signs or symptoms that impact patient performance status

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Body mass index ≤ 35
* No concurrent uncontrolled illness including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Ventricular arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements
* No uncontrolled chest or abdominal pain
* No oral or facial pain exacerbated by an oral device
* No stress incontinence
* No COPD, interstitial lung disease, pulmonary embolism, or hemorrhage within the past 6 months
* No history of pulmonary fibrosis or pulmonary hypertension
* No oxygen requirement at baseline
* No asthma
* No occupational lung disease, including, but not limited to, asbestos exposure
* No polycythemia
* No history of connective tissue disease

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the lung
* At least 6 months since prior lung surgery
* No prior amiodarone hydrochloride
* No prior high-dose chemotherapy with autologous or allogeneic hematopoietic stem cell transplantation
* No concurrent combination antiretroviral therapy for HIV-positive patients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-05; Primary Completion 2012-08-23 (Actual); Study Completion 2012-08-23 (Actual)

PRIMARY OUTCOMES:
DLCO, FVC, and FEV1 as measured by pulmonary function testing | Prior to participation in a Phase I trial

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N. Vaishampayan, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials